CLINICAL TRIAL: NCT05488691
Title: What Works and Why? Eye Movement Desensitization and Reprocessing as a Potential Treatment for Substance Use Disorders
Brief Title: Eye Movement Desensitization and Reprocessing as a Treatment for Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Hugo López-Pelayo, Interim Junior Group Leader, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI20/00506
Record Dates: First submitted 2022-06-02; First posted 2022-08-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eye Movement Desensitization and Reprocessing therapy (Experimental): 8 to 10 individual 60-minutes sessions over 2 months.
  Interventions: Behavioral: EMDR; Behavioral: TAU
- Treatment as usual (Active Comparator): Same periodicity as the experimental group and at the same time range.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: EMDR — The first session consists of recording the patient's history. In the second session the therapist evaluates the presence of coping mechanisms of the patient and, if necessary, suggests extra coping techniques. The following sessions are devoted to the reprocessing process. During these sessions, a target memory is identified and processed using EMDR. After a total of 8-10 sessions, it is expected that the patient will have achieved physiological reconciliation, relieved distress, and the ability to reformulate negative beliefs.
  Arms: Eye Movement Desensitization and Reprocessing therapy
Behavioral: TAU — treatment as usual for substance use disorders

SUMMARY:
Substance Use Disorders (SUD) are often comorbid with psychological trauma, however, the complex interaction between the two is not yet fully understood. Most addiction-specialized professionals do not engage in exploring past traumatic experiences of the patients due to personal, professional, and educational barriers. Therefore, psychological trauma remains highly undetected and its contribution to the development and maintenance of SUD is neglected. This compromises the therapeutic results of most interventions, with relapse rates in SUD still remaining impressively high. EMDR is one of the most effective interventions for Post-Traumatic Stress Disorder (PTSD), and has been applied to other disorders that are often comorbid with trauma, such as psychosis and depression, with promising results. Nevertheless, its application in SUD is still limited. Taken altogether, there is a need to clarify the efficacy of Eye Movement Desensitization and Reprocessing (EMDR) therapy in SUD, as well as the mechanisms of action that mediate its potential therapeutic effects.

The aim of this study is to 1) determine the efficacy of EMDR therapy in patients with SUD comorbid with psychological trauma, as well as whether changes in these clinical variables correspond to changes in salivary cortisol levels- a robust marker of the Hypothalamic-Pituitary-Adrenal (HPA) axis; 2) investigate the mechanisms of action of EMDR therapy, paying special attention to the key role that the cerebellum might play in mediating its therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-5 diagnosis of moderate to severe SUD, assessed by a clinical interview.
* No active drug consumption.
* Having experienced one or more traumatic events, assessed by the Life Event Checklist DSM-5 (LEC-5) and the Childhood Trauma Questionnaire (CTQ).
* Current posttraumatic symptoms, evaluated with the Impact Event Scale-Revised (IES-R).
* Aged from 18 to 65 years old.
* Sign an informed consent to participate in the study.
* Capable of speaking and comprehending Catalan or Spanish.

Exclusion Criteria:

* Having received a trauma-focused therapy within the last 5 years.
* Severe dissociative symptoms according to the Dissociative Experience Scale (DES).
* Presence of acute suicidal ideation.
* Acute episode of a comorbid psychiatric disorder.
* Severe cognitive impairments.
* Medical illness that compromises the HPA-axis.
* Long-term exposure to corticoids.
* Claustrophobia.
* Subjects with pacemakers.
* Presence of metallic objects within the body.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
time to relapse | 2 months
  Relapse is defined as a return to the addictive behavior, different from a punctual consumption, which is considered as a lapse. This will bee measured by the Time Line Follow Back self-report (TLFB)

SECONDARY OUTCOMES:
changes in functional connectivity | 2 months
  measured by resting-state fMRI
percentage of conditioned eyeblink responses (CR) | 2 months
  measured by the Eyeblink Conditioning System
CR latency, CR onset, and CR amplitude. | 2 months
  measured by the Eyeblink Conditioning System
Hair and salivary cortisol levels | 2 months
  Comparison of the Area Under the Curve pre and post treatment
Craving | 2 months 3 months and 5 months
  Self-report measurement
Total amount of substance consumed during the previous month | 2 months, 3 months and 5 months
  measured by the TLFB
Changes in depressive symptomatology | 2 months, 3 months and 5 months
  measured by Beck's Depression Inventory (BDI)
Changes in anxious symptomatology | 2 months, 3 months and 5 months
  measured by The State-Trait Anxiety Inventory (STAI)
Changes in posttraumatic symptomatology | 2 months, 3 months and 5 months
  measured by Clinician-Administered PTSD Scale (CAPS)
Changes in global functioning | 2 months, 3 months and 5 months
  measured by Functioning Assessment Short Test (FAST)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez DF, Blithikioti C, Piazza F, Nuno L, Blanco L, Rodriguez-Rey A, Munoz-Moreno E, Balcells-Olivero M, Miquel L. Eye movement desensitisation and reprocessing as a potential treatment for substance use disorders: study protocol. Eur J Psychotraumatol. 2025 Dec;16(1):2531595. doi: 10.1080/20008066.2025.2531595. Epub 2025 Aug 12. PMID 40792354